CLINICAL TRIAL: NCT02532426
Title: Influence of Chronic Hypoxia on Oxidative Phenotype in Patients With Chronic Obstructive Pulmonary Disease
Acronym: OXYPHEN
Status: Terminated | Type: Observational
Why Stopped: Lack of inclusion
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: SYNAPSE assocation (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1108100; 2011-A00856-35 (Other: AFSSAPS)
Record Dates: First submitted 2015-08-21; First posted 2015-08-25 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; Muscle biopsy; Chronic hypoxia; OXYPHEN; Oxydative phenotype; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD patients with chronic hypoxemia: COPD patients with chronic and severe arterial hypoxemia at rest (paO2<55mmHg).
  Interventions: Procedure: Muscle biopsy
- COPD patients with normoxia: COPD patients with normoxia at rest (paO2>67mmHg), matched for age, sex, bronchial obstruction and lean mass.
  Interventions: Procedure: Muscle biopsy

INTERVENTIONS:
Procedure: Muscle biopsy — The biopsy is performed on the vastus lateralis muscle at rest and 2 hours after an acute exercise, with a local anesthesia.

SUMMARY:
In addition to chronic airflow obstruction, patients with Chronic Obstructive Pulmonary Disease (COPD) suffer from skeletal muscle dysfunction which is a prominent and disabling feature and also an independent determinant of survival. Muscular impairment involves loss of muscle oxidative phenotype (OXPHEN: a slow-to-fast shift in fibre types and reduced oxidative capacity). Since hypoxia obviously is a key feature of COPD, the aim of this study is to elucidate the role of hypoxia in loss of muscle OXPHEN.

Thus, OXPHEN and expression levels of its key regulators will be determined in the baseline biopsies for association with the degree of hypoxemia. In addition, expression levels of the key OXPHEN regulators will be measured in pre/post exercise biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD confirmed according to GOLD score.
* Hypoxemia group: resting arterial paO2 <55 mmHg.
* Normoxemia group : resting arterial paO2 > 67 mmHg

Exclusion Criteria:

* Unstable cardiorespiratory status (acute respiratory failure)
* Oxygen treatment started
* Inclusion in a pulmonary rehabilitation program in the last 6 months
* Anticoagulant treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients with chronic hypoxemia and with normoxemia
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2012-05-18 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Level of expression of muscle messenger ribonucleic acid (mRNA) of HIF-1α and PGC-1α | Day 1
  Comparison of expression levels of Hypoxia-inducible Factors (HIF-1α) and Peroxisome proliferator-activated receptor gamma, coactivator 1 alpha (PGC-1α), two OXYPHEN regulators, in muscle biopsy, between COPD patients with chronic hypoxemia and those with normoxemia

SECONDARY OUTCOMES:
Type I muscle fibers | Day 1
  It is an indicator of the muscle phenotype (with a muscle biopsy). It used to compared the muscle phenotype in the 2 groups of patients. It is a percentage.
Oxidative enzyme capacity | Day 1
  It is an other indicator of the muscle phenotype (with a muscle biopsy). It used to compared the muscle phenotype in the 2 groups of patients.
Level of expression of muscle mRNA of HIF-1α after acute exercise | Day 1
  Comparison of response to acute exercise for expression level of HIF-1α (an OXYPHEN regulator) in muscle biopsy between the 2 groups.
Level of expression of muscle mRNA of PGC-1α after acute exercise | Day 1
  Comparison of response to acute exercise for expression level of PGC-1α (an OXYPHEN regulator) in muscle biopsy between the 2 groups.

CONTACTS AND LOCATIONS:
Overall Officials: COSTES Frédéric, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No